CLINICAL TRIAL: NCT03057847
Title: Management of Hepatitis C Virus (HCV) Infection in Pregnant Women With Opioid Use Disorder (OUD): the Potential of an Integrated Medical Home Model: Phase IV Trial of Sofosbuvir/Velpatasvir (SOF/VEL) in Postpartum Women With Chronic HCV
Brief Title: Sofosbuvir/Velpatasvir in Postpartum Women With Opioid Use Disorder and Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elizabeth Krans, MD (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Krans, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19030088
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C, Chronic; Opioid-use Disorder
MeSH Terms: conditions — Hepatitis C, Chronic; Opioid-Related Disorders | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SOF/VEL (Experimental): Sofosbuvir/Velpatasvir, One tablet (400 mg of sofosbuvir and 100 mg of velpatasvir) taken orally once daily for 12 weeks in the postpartum period
  Interventions: Drug: Sofosbuvir/Velpatasvir

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir — Sofosbuvir/Velpatasvir One tablet (400 mg of sofosbuvir and 100 mg of velpatasvir) taken orally once daily for 12 weeks in the postpartum period
  Other Names: Epclusa

SUMMARY:
Incorporating Hepatitis C Virus (HCV) treatment into opioid maintenance treatment program clinical protocols is an innovative health care delivery model that has been associated with improved HCV treatment uptake in non-pregnant, drug-using populations. This "medical home" approach would combine HCV and opioid maintenance treatment into one treatment regimen and incorporate the expertise of obstetricians, hepatologists, substance abuse treatment providers and pediatricians into one comprehensive clinical care model. The purpose of this study is to evaluate the feasibility/acceptability of a combined, peripartum HCV and opioid maintenance treatment program on adherence to HCV treatment regimens and evaluate the rate of intravenous drug use (IVDU) recidivism, HCV reinfection and health related Quality of Life (QOL) in women with opioid use disorder (OUD) during the first postpartum year.

The protocol involves three separate study phases. All 3 study phases will occur with support from hepatology providers at Magee-Womens Hospital. Phase 1 involves screening, enrollment and a baseline assessment of liver function, HCV infection (genotype, viral load) and blood and urine studies in HCV-infected patients during pregnancy. In Phase 2, subjects will undergo 12 weeks of sofosbuvir/velpatasvir therapy initiated at 2 weeks postpartum. Feasibility/acceptability and adherence to sofosbuvir/velpatasvir will be assessed at 4, 8 and 12 weeks of therapy. In Phase 3, subjects will continue to be followed for 15 months after treatment completion. Treatment effectiveness and sustained virologic response (SVR) will be evaluated at 3 months and rates of IVDU recidivism, HCV reinfection and patient centered outcomes such as health related quality of life (QOL) will be assessed at 6, 9 and 12 months following treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Able and willing to provide written informed consent to be screened for and take part in the study procedures
3. Able and willing to provide adequate contact information
4. Chronic Hepatitis C Virus (HCV), genotype 1 (1a, 1b), 2 (2a, 2b), 3, 4, 5, 6 infection, defined as a HCV antibody and detectable HCV ribonucleic acid (RNA) viral load at screening
5. Pregnancy at 28 + 0 to 37 + 6 weeks' gestation at enrollment with gestational dating confirmed by ultrasound
6. Documented negative Hepatitis B testing within 3 months prior to enrollment
7. Negative human immunodeficiency virus (HIV) testing within 3 months prior to enrollment
8. Per participant report at screening and enrollment, agrees not to participate in other research studies involving drugs or medical devices for the duration of study participation
9. Plans to deliver at Magee-Womens Hospital of University of Pittsburgh Medical Center (UPMC)

Exclusion Criteria:

1. Participant report of any of the following at Screening or Enrollment:

   1. Previous treatment for Hepatitis C virus with a sofosbuvir based regimen
   2. Use of any medications contraindicated with concurrent use of sofosbuvir/velpatasvir according to the EPCLUSA package insert
   3. Plans to relocate away from the study site area in the next 18 months
   4. Current sexual partner is known to be infected with HIV or Hepatitis B virus
   5. History of decompensated cirrhosis (history of variceal bleed, ascites or hepatic encephalopathy)
2. Reports participating in any other research study involving drugs or medical devices within 60 days or less prior to enrollment
3. Ongoing illicit drug use evidenced by positive urine drug screen with appropriate confirmatory testing for anything other than marijuana since the first prenatal visit that cannot be explained by a prescribed medication
4. Breastfeeding or pumping and feeding infant breastmilk
5. At screening or enrollment, as determined by the Protocol Chair, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease (other than Hepatitis C)
6. Has any of the following laboratory abnormalities at Screening:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 10 times the upper limited of normal
   2. Hemoglobin less than 10 g/dL
   3. Platelet count less than 90,000 per mm3
   4. International normalized ratio (INR) > 1.5
   5. Glomerular filtration rate (GFR) < 40
7. Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Krans, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOF/VEL
Started | 32
Treatment Initiation | 21
Completed | 16
Not Completed | 16
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Arm/Group | SOF/VEL
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.88 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Initiating in Hepatitis C Virus (HCV) Treatment
Description: Number of participants initiating HCV treatment
Time Frame: Delivery to 10 months postpartum
Population: Number of participants initiating HCV treatment
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 32
Participants | 21

2. Secondary Outcome: Intravenous Drug Use Recidivism
Description: Rate of intravenous drug use recidivism by participant self-report and Urine Drug Screening
Time Frame: 15 months post-treatment, up to 18 months
Population: Rate of intravenous drug use recidivism by participant self-report and Urine Drug Screening
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 16
Participants | 3

3. Secondary Outcome: HCV Reinfection
Description: Count of participants 15 months post-treatment with Hepatitis C Virus reinfection as measured by related lab tests
Time Frame: 15 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 16
Participants | 0

4. Secondary Outcome: Health-related Quality of Life
Description: Health-related quality of life using Promise 57 scale
Time Frame: 15 months post-treatment
Population: Data was not collected and will not be reported due to lack of survey development
Arm/Group | SOF/VEL
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Achieving Sustained Virologic Response (SVR)
Description: Number of participants with non-detectable Hepatitis C Virus (HCV) Ribonucleic acid (RNA) post-treatment as measured by SVR testing
Time Frame: End of treatment (12 weeks postpartum) up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 13
Participants | 13

6. Secondary Outcome: Number of Participants Reporting Treatment Side Effects
Description: Number of participants reporting treatment side effects using standardized list
Time Frame: End of treatment (12 weeks postpartum)
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 21
Participants | 12

7. Secondary Outcome: Number of Missed Treatment Doses
Description: Treatment adherence assessed by missed treatment doses
Time Frame: End of treatment (12 weeks postpartum)
Measure: Median (95% Confidence Interval); unit: doses
Units Other Than Participants: doses of treatment medication
Arm/Group | SOF/VEL
Number analyzed (Participants) | 16
Number analyzed (doses of treatment medication) | 84
doses | 2 [0 to 5]

ADVERSE EVENTS:
Time Frame: Treatment Initiation, up to 18 months
Arm/Group | SOF/VEL
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 12/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOF/VEL (N=32)
Headaches (Nervous system disorders) | 12 (44)
Fatigue (General disorders) | 7 (22)
Nausea (Gastrointestinal disorders) | 3 (19)
Insomnia (Psychiatric disorders) | 2 (5)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood in Stool (General disorders) | 1 (1)
Teeth sensitivity (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Due to lower than expected enrollment numbers and thus, insufficient power for multivariable analytic approaches, we were unable to perform the analyses originally proposed for this study. Thus, we had to adjust our statistical analysis plan to fit the number of participants actually enrolled in the study which now consists of largely descriptive and bivariate statistics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03057847/Prot_SAP_000.pdf